CLINICAL TRIAL: NCT06532929
Title: Safety and Clinical Performance Assessment of Sport Surgery Products - A Post-market Clinical Follow-up
Brief Title: Sport Surgery Products Outcomes - A Post-market Follow-up
Status: Recruiting | Type: Observational
Sponsor: Teknimed (Industry)
Responsible Party: Sponsor
Other Study IDs: SM01-TK-SPORTS
Record Dates: First submitted 2024-07-25; First posted 2024-08-01 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Sport Surgery
Keywords: knee; shoulder; sport; surgery; suture; ligamentoplasty; anchors; screw; resorbable; pins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- EUROSCREW NG PLA knee (ACL) surgery: Patients included for anterior crucial ligament of knee surgery with EUROSCREW NG PLA
  Interventions: Device: Orthopaedic surgeries (knee)
- EUROSCREW NG PLA knee (PCL) surgery: Patients included for posterior crucial ligament of knee surgery with EUROSCREW NG PLA
  Interventions: Device: Orthopaedic surgeries (knee)
- EUROSCREW NG PLA ankle surgery: Patients included for ankle surgery with EUROSCREW NG PLA
  Interventions: Device: Orthopaedic surgeries (ankle)
- EUROSCREW NG PLA/TCP knee (ACL) surgery: Patients included for anterior crucial ligament of knee surgery with EUROSCREW NG PLA/TCP
  Interventions: Device: Orthopaedic surgeries (knee)
- EUROSCREW NG PLA/TCP knee (PCL) surgery: Patients included for posterior crucial ligament of knee surgery with EUROSCREW NG PLA/TCP
  Interventions: Device: Orthopaedic surgeries (knee)
- ISOFIX knee (ACL) surgery: Patients included for anterior crucial ligament of knee surgery with ISOFIX
  Interventions: Device: Orthopaedic surgeries (knee)
- A'LINK'S shoulder surgery: Patients included for shoulder surgery with A'LINK'S
  Interventions: Device: Orthopaedic surgeries (shoulder)
- SUTUR'LINK surgery: Patients included for surgery with SUTUR'LINK
  Interventions: Device: Orthopaedic surgeries
- PINS foot surgery: Patients included for foot surgery with PINS
  Interventions: Device: Orthopaedic surgeries (foot)

INTERVENTIONS:
Device: Orthopaedic surgeries (ankle) — ankle lateral ligament reconstruction in ligamentoplasty procedures
  Groups: EUROSCREW NG PLA ankle surgery
Device: Orthopaedic surgeries (shoulder) — rotator cuff repair
  Groups: A'LINK'S shoulder surgery
Device: Orthopaedic surgeries (knee) — knee cruciate ligaments reconstruction in ligamentoplasty procedures
  Groups: EUROSCREW NG PLA knee (ACL) surgery; EUROSCREW NG PLA knee (PCL) surgery; EUROSCREW NG PLA/TCP knee (ACL) surgery; EUROSCREW NG PLA/TCP knee (PCL) surgery; ISOFIX knee (ACL) surgery
Device: Orthopaedic surgeries — rotator cuff repair or closure of capsule after arthroplasty surgery
  Groups: SUTUR'LINK surgery
Device: Orthopaedic surgeries (foot) — stabilization of metatarsal and phalangeal osteotomies during treatment of hallux
  Groups: PINS foot surgery

SUMMARY:
Teknimed is currently conducting a post-market clinical follow-up which will confirm performance, safety and usability for all the Teknimed range of Sports products. TEKNIMED has developed several devices currently used in orthopaedic surgery. With the increasing use of these procedures, there is a need for real-life long-term safety and efficacy data on these products.

The study is a retrospective and prospective global, single arm, non-controlled, multicentric, ambispective observational study. Patients will be followed as per local standard medical care of the site.

DETAILED DESCRIPTION:
It is admitted that:

* Bioabsorbable interference screws are frequently used for graft attachment in knee cruciate ligament reconstruction,
* Bioabsorbable pins are indicated for the realignment and fixation of epiphyseal fractures, osteotomies, arthrodesis and bone grafts of toes,
* Non-absorbable suture is usually used for the repair and the reinforcement of ligaments or tendons structures during surgery procedures,
* Anchor devices are usually used for the repair of rotator cuff tendons and biceps tenodesis.

Furthermore, resorption properties of many available devices (screws, pins) that are marketed as bioabsorbable may be different and not always very well defined.

This retro-prospective study is performed to confirm the safety and performance of TEKNIMED sports surgery products in their current clinical use.

Studied products include - but are not restricted to - the following TEKNIMED products:

* EUROSCREW® NG
* ISOFIX®
* SUTUR'LINK®
* A'LINK'S®
* BIORESORBABLE PINS

And following associated TEKNIMED instrumentation:

* ACL Instrumentation
* A'LINK'S® Instrumentation
* STAINLESS STEEL PINS

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older.
* Be willing to sign an informed consent approved by IRB or EC (where applicable) or not being opposed to the use of their clinical data in the study (France)

For prospective inclusion:

- Be considered for a surgery with one of the TEKNIMED sports surgery product comprised in this study.

For retrospective inclusion:

* Have undergone a surgery with a TEKNIMED sports surgery product between the 1st January 2016 and the date of the site initiation visit.
* Be informed of the study and not being opposed to the use of their clinical data in the study (France) or be willing to sign an informed consent during the first follow-up visit following the site initiation (when applicable).

Exclusion Criteria:

* Patients presenting one of the following conditions will not be included: under trusteeship or guardianship, pregnancy
* Anyone of the contraindications mentioned in the respective IFU of each device under study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People suffering from tears or ruptures of ligaments or tendons and in need of an orthopaedic surgery, according to the specific intended uses related to each device.
Sampling Method: Non-Probability Sample
Enrollment: 390 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2036-11 (Estimated); Study Completion 2036-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of join function | 4 years (until the lifetime of the device)
  Function will be evaluated from standardized and validated clinical questionnaires, with few questions relative to domains such as pain, mobility, range of motion... which are specific for one joint
Adverse event | 5 years
  Adverse event related to sports surgery products

SECONDARY OUTCOMES:
Pain level | 4 years
  Pain evaluated by Visual Analogue Scale (VAS): on a scale of 0 to 10, with 0 being no pain and 10 being the most severe pain at the Baseline and at the Follow-up visits
Antalgic consumption | 4 years
  Antalgic consumption and the drug type at the Baseline and at the Follow-up visits
Patients' satisfaction | 4 years
  Patient satisfaction assessed using a 3-question patient satisfaction questionnaire (Yes/No/Without opinion) at the Follow-up visits
Quality of patient life | 4 years
  Quality of patient life assessed using Well-Being questionnaire (6 questions with a scale of 0 to 10, with 0 being not at all and 10 being the better response at the Baseline and at the Follow-up visits)
Radiological outcomes | 4 years
  Evaluation of implants integrity/ resorption Bioresorbable screws, pins and anchors will be classified as "degraded", "partially intact" or "intact", as observed on imaging exam.
Devices and instrumentations usability | Once, during surgery
  Instrumentations usability assessed by physician evaluation of the sucessive phases of surgery.
  The physician is asked to evaluate the successive phases of the surgery to assess the global device usability. For each technical phase, he has to choose between 3 propositions: Easy, Difficult or Impossible. At the end of the surgical procedure, the surgeon is asked to assess the resulting joint stability (stable or unstable).

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Milaire, Aubenas, Ardèche
  - Centre Claude Bernard, Guilherand-Granges, Ardèche
  - Centre Mistral -Clinique Pasteur, Guilherand-Granges, Ardèche
  - Orthopole des 3 provinces, Brive-la-Gaillarde, Corrèze
  - Clinique Pasteur, Bergerac, Dordogne
  - Médipôle Toulouse, Toulouse, Haute-Garonne
  - Clinique Chénieux, Limoges, Haute-Vienne
  - Clinique St Privat, Boujan-sur-Libron, Hérault
  - Clinique Via Domitia, Lunel, Hérault
  - Clinique Esquirol Saint-Hilaire, Agen, Lot-et-Garonne

IPD SHARING:
Plan to Share IPD: No